CLINICAL TRIAL: NCT05533320
Title: Evaluation Of Benefits of The Portable Scalp Cooling System (PSCS) in Metastatic Breast Cancer Patients on Taxane-Based Chemotherapy
Brief Title: Portable Scalp Cooling System for the Improvement of Chemotherapy-Induced Hair Loss in Patients With Metastatic Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided to withdraw
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21030; NCI-2022-06837 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21030 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Supportive care (PSCS) (Experimental): Patients undergo scalp cooling using the PSCS 30 minutes before, during, and for up to 2 hours after completion of chemotherapy for 6 chemotherapy sessions.
  Interventions: Device: Cold Cap Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Device: Cold Cap Therapy — Undergo scalp cooling
  Other Names: Cold Cap; Paxman Scalp Cooling System; PSCS; Scalp Cooling; Scalp Cryotherapy; Scalp Hypothermia
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the benefits of a portable scalp cooling system (PSCS) for improving chemotherapy-induced hair loss in patients with breast cancer that has spread to other places in the body (metastatic) and are undergoing taxane-based chemotherapy. The PSCS is a new system designed to reduce chemotherapy induced hair loss. The PSCS is designed as a portable unit, allowing patients to leave the infusion center after chemotherapy is completed and finish scalp cooling at home. PSCS may help improve chemotherapy-induced hair loss in patients with metastatic breast cancer receiving chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Measure efficacy of scalp cooling for patients undergoing taxane based chemotherapy for metastatic breast cancer.

SECONDARY OBJECTIVES:

I. Assess safety of PSCS in treating patients with metastatic breast cancer. II. Assess burden on nurses and infusion center team of patients using the PSCS.

III. Assess tolerability of PSCS. IV. Assess hair loss and recovery as assessed by the patient. V. Assess patient quality of life and satisfaction with treatment.

OUTLINE:

Patients undergo scalp cooling using the PSCS 30 minutes before, during, and for up to 2 hours after completion of chemotherapy for 6 chemotherapy sessions.

After completion of study, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Ability to read and understand English or Spanish for questionnaires
* Documented diagnosis of metastatic breast cancer with at least a 6 month life expectancy
* A planned course of taxane based chemotherapy in the metastatic setting, including paclitaxel, docetaxel or abraxane
* At least 6 months from the last chemotherapy causing hair loss with complete recovery of hair
* Willing to be contacted for brief annual assessments for five years
* Women of childbearing potential (WOCBP): negative urine pregnancy test
* Agreement by females of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Autoimmune disease affecting hair; e.g. alopecia areata, systemic lupus with associated hair loss
* A history of whole brain radiation with persistent hair thinning or alopecia, or concurrent whole brain radiation therapy
* Exposure to other investigational agents, drugs, device or procedure that may cause hair loss
* Patients with female pattern baldness resembling picture I-3 or higher on the Savin scale
* Any cutaneous scalp metastases
* Clinically significant liver dysfunction considered significant as determined by treating physician that would limit the patient's ability to administer the scalp cooling device
* Clinically significant renal dysfunction considered significant as determined by treating physician that would limit the patient's ability to administer the scalp cooling device
* A history of persistent grade 2 (or higher) alopecia induced by prior chemotherapeutic regimens
* Evidence of untreated or poorly controlled hyper or hypothyroidism
* American Society of Anesthesiologist Class >= 3
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Pregnant or breastfeeding
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2022-12-14 (Estimated); Primary Completion 2023-11-14 (Estimated); Study Completion 2023-11-14 (Estimated)

PRIMARY OUTCOMES:
Success in hair preservation | At 4 weeks after completion of the 6th chemotherapy cycle
  Hair loss will be measured by the patient according to the Dean Score. (Grade 0: no hair loss, grade 1: > 0 - 25%; grade 2: > 25 - 50%; grade 3: > 50 - 75%; grade 4: > 75%). Hair preservation was defined as hair loss no more than grade 2.

SECONDARY OUTCOMES:
Incidence of adverse events of PSCS | At 4 weeks, 3 months, and 6 months following the conclusion of 6 cycles of chemotherapy
  Will be determined by spontaneous reporting of adverse events and negative scalp changes determined by physical examination. Frequency tables will be used to summarize these events.
Burden on nurses and infusion center team | Up to 1 year
  The workload impact will be assessed via surveys distributed to nurses, and descriptive analysis will be used to explore the collected data.
Tolerability of PSCS | Up to 1 year
  Will be determined by the proportion of patients who completed all planned cycles of chemotherapy using the PSCS will be assessed (including 95% CI).
Hair loss recovery | Up to 1 year
  Patient self-assessment of hair loss at each chemotherapy infusion.
Patients quality of life | Up to 30 days after the last dose of treatment
  Will be measured by EORTC-QLQ-30 quality of life questionnaire. Changes will be summarized descriptively and comparison with baseline will be carried out using paired t-test (or non-parametric paired test when suitable). In addition, repeated measures one-way ANOVA will also be used where appropriate to evaluate changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: James R Waisman, Principal Investigator — City of Hope Medical Center